CLINICAL TRIAL: NCT04123028
Title: The Association Between Blood Eosinophils and Clinical Outcomes of Chronic Obstructive Pulmonary Disease Patients: A Prospective Study
Brief Title: The Association Between Blood Eosinophilsp in Thai COPD Patients: A Prospective Study
Status: Completed | Type: Observational
Sponsor: Prince of Songkla University (Other)
Responsible Party: Principal Investigator, Siwasak Juthong, Faculty of Medicine, Prince of Songkla University
Other Study IDs: 60-319-14-3
Record Dates: First submitted 2019-10-08; First posted 2019-10-10 (Actual); Last update posted 2019-10-11 (Actual); Status verified 2019-10

CONDITIONS: Copd
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- eosinophilic COPD patient: COPD patient with blood eosinophil equal or > 300 cells/µL
  Interventions: Other: observatory
- non-eosinophilic COPD patient: COPD patient with blood eosinophil < 300 cells/µL
  Interventions: Other: observatory

INTERVENTIONS:
Other: observatory — observation for 1 year period
  Other Names: clinical outcomes

SUMMARY:
The association of blood eosinophil as a biomarker for eosinophilic Thai COPD patients, such as COPD exacerbation, hospital admission, lung functions and mortlity.

DETAILED DESCRIPTION:
The prospective one year study in Thai COPD patients for the clinical outcomes of COPD compare between eosinophilic and non-eosinophilic which determine by blood eosinophil counts equal or more than 300 cells/microliters. The primary outcomes was COPD exacerbation, the secondary outcomes were lung function, dyspnea and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of COPD by GOLD criteria

Exclusion Criteria:

1. high blood eosinophil from known causes such as systemic corticosteroid use, malignancy, parasitic infection
2. Patients who had previous acute exacerbation within 30-day before study entry
3. Patients who had previous systemic corticosteroids used within 30-day before study entry

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Thai COPD patients in out-patient department
Sampling Method: Non-Probability Sample
Enrollment: 145 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Acute worsening of respiratory symptoms | 1 year
  acute severe worsening of respiratory symptoms

SECONDARY OUTCOMES:
Physiological outcomes | 1 year
  Forced expiratory volume in one second
health related quality of life | 1 year
  Chronic Obstructive Pulmonary Disease Assessment Test (CAT) scores which the minimum 0 and maximum 40 values, and whether higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Kanung Saejiam, MS, Study Director — Prince of Songkla University
Locations (1):
- Faculty of Medicine, Prince of Songkla university, Songkhla, Thailand

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bafadhel M, Pavord ID, Russell REK. Eosinophils in COPD: just another biomarker? Lancet Respir Med. 2017 Sep;5(9):747-759. doi: 10.1016/S2213-2600(17)30217-5. Epub 2017 Jun 7. PMID 28601554
- [Derived] Juthong S, Kaenmuang P. Association between blood eosinophils with exacerbation and patient-reported outcomes in chronic obstructive pulmonary disease patients in an endemic area for parasitic infections: a prospective study. J Thorac Dis. 2020 Sep;12(9):4868-4876. doi: 10.21037/jtd-19-4101. PMID 33145060